CLINICAL TRIAL: NCT07350616
Title: The Effect of the 5T Teach-Back Method in Respiratory Exercise and Incentive Spirometer Training on Knowledge Level, Practical Skills, Respiratory Parameters, and Patient Satisfaction: A Randomized Controlled Study
Brief Title: The Effect of the 5T Teach-Back Method on Respiratory Exercise and Incentive Spirometer Training
Acronym: TEACH-BREATHE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Cigdem Erdem, Assistant Professor, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 973-973-11
Record Dates: First submitted 2025-12-28; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pulmonary Complications; Atelectasis; Patient Education; Respiratory Exercises; Incentive Spirometry
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5T Teach-Back Education Group (Experimental): Participants receive preoperative respiratory exercise and incentive spirometer training using the 5T Teach-Back method.
  Interventions: Behavioral: 5T Teach-Back-Based Respiratory Exercise and Incentive Spirometer Education
- Standard Education Group (Active Comparator): Participants receive routine verbal education on respiratory exercises and incentive spirometer use provided by clinical nurses.
  Interventions: Behavioral: Standard Verbal Respiratory Education

INTERVENTIONS:
Behavioral: 5T Teach-Back-Based Respiratory Exercise and Incentive Spirometer Education — This intervention involves preoperative respiratory exercise and incentive spirometer education delivered using the structured 5T Teach-Back method. Education is provided individually by a trained nurse and includes demonstration, patient return demonstration, and repeated instruction until correct understanding and performance are achieved. The five steps of the 5T Teach-Back approach (Triage, Tools, Take Responsibility, Tell Me, and Try Again) are systematically applied to ensure patient comprehension and skill mastery. Sessions last approximately 20-30 minutes and are completed before surgery. Unlike routine verbal education, this intervention actively engages patients in explaining and performing the exercises in their own words, allowing immediate correction of misunderstandings and reinforcing correct technique
  Arms: 5T Teach-Back Education Group
Behavioral: Standard Verbal Respiratory Education — This intervention consists of routine verbal education on respiratory exercises and incentive spirometer use provided by clinical nurses as part of standard preoperative care. Education is delivered according to usual clinical practice without a structured teaching framework, return demonstration, or formal assessment of patient understanding. No standardized duration, repetition, or feedback process is applied. This intervention reflects typical routine care and differs from structured educational approaches by relying solely on conventional verbal instruction.
  Arms: Standard Education Group

SUMMARY:
Breathing problems after surgery are common and can lead to serious complications such as low oxygen levels, lung collapse, or pulmonary embolism. These problems increase patient risk and place an additional burden on the healthcare system. Breathing exercises and incentive spirometer use are important methods to prevent these complications. However, many patients have difficulty understanding and correctly performing these exercises when education is limited to standard verbal instructions. This randomized controlled study aims to evaluate whether the 5T Teach-Back education method improves patients' understanding, practical skills, respiratory outcomes, and satisfaction compared with standard verbal education. The study will be conducted in a university hospital and will include 76 adult patients undergoing abdominal surgery under general anesthesia. Participants will be randomly assigned to either an intervention group or a control group.

Patients in the intervention group will receive preoperative breathing exercise and incentive spirometer training using the 5T Teach-Back method, which encourages patients to explain the information back in their own words and repeat the skills until they are correctly understood. Patients in the control group will receive routine verbal education provided by clinical nurses. Outcomes will be measured before surgery and again within 24-72 hours after surgery. These outcomes include patients' knowledge level, correct performance of breathing exercises and spirometer use, respiratory rate, oxygen saturation, lung function test results, and patient satisfaction with nursing care. The results of this study are expected to show whether the 5T Teach-Back method is more effective than standard education in improving postoperative respiratory care and patient satisfaction. The findings may help standardize patient education practices and support nurses in delivering more effective respiratory training before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Scheduled for abdominal surgery under general anesthesia
* Postoperative use of respiratory exercises and incentive spirometry is recommended
* Expected postoperative hospital stay of more than 3 days
* Able to read and write and able to communicate effectively
* Conscious, cooperative, and oriented
* Willing to participate voluntarily and able to provide written informed consent

Exclusion Criteria:

* Severe neurological or cognitive impairment
* Unstable vital signs or hemodynamic instability
* Anticipated or required postoperative intensive care unit admission
* Severe pain that prevents participation in education or assessments
* Visual or communication impairments that limit participation in education

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Patient Knowledge and Correct Performance of Respiratory Exercises and Incentive Spirometer Use | From baseline (preoperative period) to 24-72 hours postoperatively
  Patient knowledge and correct performance of respiratory exercises and incentive spirometer use will be assessed using a structured knowledge test and observation-based checklists. Knowledge level will be evaluated with a short multiple-item test, and performance accuracy will be assessed by direct observation of breathing exercises and incentive spirometer use. Higher scores indicate better understanding and correct application of the techniques.

SECONDARY OUTCOMES:
Pulmonary Function Test | 24-72 hours postoperatively
  Pulmonary function will be assessed postoperatively using spirometry. The primary parameter will be the FEV1/FVC ratio (%), where higher values indicate better pulmonary function.
Patient Satisfaction | 24-72 hours postoperatively
  Patient satisfaction will be assessed using the Newcastle Satisfaction with Nursing Scales (NSNS). The NSNS was originally developed by Thomas et al. (1996) to evaluate patients' experiences and satisfaction with nursing care and was adapted and validated in Turkish by Akın and Erdoğan (2007). The scale consists of 19 items rated on a 5-point Likert scale. Item scores are summed and transformed to yield a total satisfaction score ranging from 0 to 100. Higher scores indicate greater satisfaction with nursing care, with a score of 100 representing the highest possible level of satisfaction.
Respiratory Parameter (SpO₂) | From baseline (preoperative period) to 24-72 hours postoperatively
  Peripheral oxygen saturation (SpO₂, %) will be measured pulse oximetry. Changes between baseline (preoperative) and postoperative assessment will be compared between study group
Respiratory Rate | From baseline (preoperative period) to 24-72 hours postoperatively
  Respiratory rate (breaths/min) will be measured using routine clinical assessment. Changes between baseline (preoperative period) and postoperative assessment will be compared between study groups.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang J, Hu H, Sun J, Zhang Q, Chen Z, Wang Q, Zhu M, Yao J, Yuan H, Zhang X. The effectiveness of health education based on the 5Ts for teach-back on oral nutritional supplements compliance of post-discharge patients after surgery for gastric cancer: a randomized controlled trial. Support Care Cancer. 2023 Feb 11;31(3):157. doi: 10.1007/s00520-023-07581-1. PMID 36773116
- [Background] Anderson KM, Leister S, De Rego R. The 5Ts for Teach Back: An Operational Definition for Teach-Back Training. Health Lit Res Pract. 2020 Apr 9;4(2):e94-e103. doi: 10.3928/24748307-20200318-01. PMID 32293689